CLINICAL TRIAL: NCT02650414
Title: Pilot Study of Autologous Anti-CD22 Chimeric Antigen Receptor Redirected T Cells in Pediatric Patients With Chemotherapy Resistant Or Refractory Acute Lymphoblastic Leukemia
Brief Title: CD22 Redirected Autologous T Cells for ALL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15CT055; 15-012219; 823312
Record Dates: First submitted 2015-12-22; First posted 2016-01-08 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: B Cell Leukemias; B Cell Lymphomas
Keywords: Biological: CART 22
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pediatric patients with relapsed or refractory B-cell acute lymphoblastic leukemia (Experimental)
  Interventions: Biological: Cohort 1; Biological: Cohorts 2; Biological: Cohort 3

INTERVENTIONS:
Biological: Cohort 1 — Subjects <50kg will receive 0.2-1 x 10^7 CART22 cells/kg as a split dose over three days as follows:
  Day 1, 10% fraction: 0.2-1x10^6 CART22 cells/kg Day 2, 30% fraction: 0.6-3x10^6 CART22 cells/kg Day 3, 60% fraction: 1.2-6x10^6 CART22 cells/kg
  Subjects ≥50kg will receive 1-5x10^8 CART22 cells as a split dose over three days as follows:
  Day 1, 10% fraction: 1-5x10^7 CART22 cells/kg Day 2, 30% fraction: 0.3-1.5x10^8 CART22 cells/kg Day 3, 60% fraction: 0.6-3x10^8 CART22 cells/kg
Biological: Cohorts 2 — Subjects <50kg will receive 0.2-1 x 10^7 CART22-65s cells/kg as a split dose over three days as follows:
  Day 1, 10% fraction: 0.2-1x10^6 CART22-65s cells/kg Day 2, 30% fraction: 0.6-3x10^6 CART22-65s cells/kg Day 3, 60% fraction: 1.2-6x10^6 CART22-65s cells/kg
  Subjects ≥50kg will receive 1-5x10^8 CART22-65s cells as a split dose over three days as follows:
  Day 1, 10% fraction: 1-5x10^7 CART22-65s cells/kg Day 2, 30% fraction: 0.3-1.5x10^8 CART22-65s cells/kg Day 3, 60% fraction: 0.6-3x10^8 CART22-65s cells/kg
Biological: Cohort 3 — Subjects <50kg will receive 0.2-1 x 10^7 CART22-65s cells as a split dose over two days as follows:
  Day 1, 25% fraction: 0.5-2.5x10^6 CAR T cells/kg Day 2, 75% fraction: 1.5-7.5x10^6 CAR T cells/kg
  Subjects ≥50kg will receive 1-5x10^8 CART22-65s cells as a split dose over two days as follows:
  Day 1, 25% fraction: 0.25-1.25x10^8 CART22-65s cells Day 2, 75% fraction: 0.75-3.75x10^8 CART22-65s cells

SUMMARY:
This is a pilot study to determine the feasibility and safety of a single dose of autologous T cells expressing CD22 chimeric antigen receptors expressing tandem TCR-ζ and 4-1BB signaling domains (CART22/CART22-65s cells) in pediatric and young adult subjects with relapsed or refractory B cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
This is a single center, single arm, dual-cohort, open-label pilot study to determine the feasibility and safety of a single dose (administered as split fractions) of autologous T cells expressing CD22 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ/4-

1BB) co-stimulatory domains (referred to as "CART22" and "CART22-65s" cells) in pediatric patients with relapsed or refractory B-cell acute lymphoblastic leukemia. Cohort assignment will be dependent on the date of consent and confirmation of eligibility by a physician-investigator as follows:

* Cohort 1: was closed to additional recruitment as of Protocol Version 8. All subjects who received CART22 cells will be retrospectively assigned to Cohort 1.
* Cohort 2: was opened as of Protocol Version 8. All subjects assigned to Cohort 2 will receive CART22-65s cells given over 3 days.
* Cohort 3: will open as of Protocol V12, with subjects enrolled sequentially after all infusion slots in Cohort 2 are filled. All subjects assigned to Cohort 3 will also receive CART22-65s cells, however the product will be administered over 2 days.

ELIGIBILITY:
1. Signed informed consent form must be obtained prior to any study procedure.
2. Relapsed or refractory B-cell ALL:

   1. 2nd or greater relapse OR
   2. Any marrow or extramedullary relapse after allogeneic HSCT and ≥ 6 months from SCT at infusion OR
   3. Any marrow relapse after CAR-modified T cell therapy OR
   4. Refractory disease defined as having not achieved a CR after > 2 chemotherapy regimens OR
   5. Patients with Ph+ ALL are eligible if they are intolerant to or have failed tyrosine kinase inhibitor therapy OR
   6. Ineligible for allogeneic SCT because of:

   i. Comorbid disease ii. Other contraindications to allogeneic SCT conditioning regimen iii. Lack of suitable donor iv. Prior SCT v. Declines allogeneic SCT as a therapeutic option after documented discussion, with expected outcomes, about the role of SCT with a BMT physician not part of the study team g. Patients with CNS3 disease will be eligible if CNS disease is responsive to therapy (at infusion, must meet criteria in Section 5.2)
3. Documentation of CD22 tumor expression in bone marrow, other tumor biopsy, CSF or peripheral blood by flow cytometry (or a recent marrow in the case of refractory disease). If the patient has received CD22-directed therapy (i.e., inotuzumab), then the marrow or other sample should be obtained after this therapy to show CD22 expression.
4. Adequate organ function defined as:

   a. A serum creatinine based on age/gender as follows:
   1. A serum creatinine based on age/gender as follows:

      Maximum Serum Creatinine (mg/dL) Age 1 to < 2 years Male 0.6 Female 0.6 Age 2 to < 6 years Male 0.8 Female 0.8 Age 6 to < 10 years Male 1.0 Female 1.0 Age 10 to < 13 years Male 1.2 Female 1.2 Age 13 to < 16 years Male 1.5 Female 1.4 Age ≥ 16 years Male 1.7 Female 1.4
   2. Adequate liver function

   i. ALT < 500 U/L ii. Bilirubin <3x upper limit of normal

   iii. ALT and/or bilirubin that exceed these ranges is acceptable if, in the opinion of the investigator (or by liver biopsy), the abnormalities are directly related to ALL infiltration of the liver

   c. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea, pulse oxygen > 92% on room air; DLCO > 40% (corrected for anemia) if PFTs are clinically appropriate as determined by the treating investigator

   d. Left Ventricle Shortening Fraction (LVSF) ≥ 28% or Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA; in cases where quantitative assessment of LVEF is not possible, a statement by the cardiologist that the ECHO shows qualitatively normal ventricular function will suffice.
5. Evidence of disease by standard morphologic or by MRD criteria. If the results of a historical biopsy (obtained at the time of the patient's most recent relapse) are available, this does not need to be repeated at screening.
6. Age 1-29 years.
7. Adequate performance status (Lansky or Karnofsky score ≥50).
8. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Active hepatitis B or active hepatitis C.
2. HIV Infection.
3. Active acute or chronic graft-versus-host disease (GVHD) requiring systemic therapy.
4. Concurrent use of systemic steroids or immunosuppressant medications. Recent or current use of inhaled steroids or physiologic replacement with hydrocortisone is not exclusionary.
5. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity.
6. Pregnant or nursing (lactating) women.
7. Receipt of a prior investigational study agent within 4 weeks prior to screening visit. *Note - patients who have received anti-CD19 CART cells (e.g., CART19/CTL019) on an investigational study where cell infusion occurred greater than 4 weeks before the screening visit are NOT excluded.

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Estimated)
Dates: Start 2016-01-13 (Actual); Primary Completion 2037-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events, including, but not limited to, cytokine release syndrome (CRS) | From date of dosing ( day 1 ) up 15 years
  grade 3 and higher toxicity rate (toxicity possibly attributed to CART22)

SECONDARY OUTCOMES:
Percentage of manufacturing products that do not meet release criteria. | 3 months
  Product must pass for vector transduction efficiency, T cell product purity, viability, sterility or due to tumor contamination.
Overall Complete Remission Rate (ORR) at Day 28. | 4 months
  Includes CR and CR with incomplete blood count recovery (CRi)
Evaluate overall response rate (CR/CRi by or at Month 6) at Month 6. | 9 months
Evaluate disease status at Month 6. | 9 months
Overall survival (OS) | 15 years
Duration of remission (DOR) | 15 Years
Number of subjects with relapse free survival (RFS) | 15 years
Number of subjects with event free survival (EFS). | 15 years
Describe cause of death (COD) when appropriate | 15 years
Describe response in terms of minimal residual disease (MRD). | 1 year
  Percentage of patients who achieve a CR associated with minimal residual disease (MRD) negative bone marrow as determined by high sensitivity flow cytometry.
Incidence of any acute GVHD | 15 year
Incidence of any grade II-IV aGVHD | 15 year
Incidence any chronic GVHD. | 15 year
Incidence any extensive, limited cGVHD. | 15 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Grupp, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Myers RM, DiNofia AM, Li Y, Diorio C, Liu H, Wertheim G, Fraietta JA, Gonzalez V, Plesa G, Siegel DL, Iannone E, Shinehouse L, Brogdon JL, Taylor C, Jadlowsky JK, Hexner EO, Engels B, Baniewicz D, Callahan C, Ruella M, Aplenc R, Barz Leahy A, McClory SE, Rheingold SR, Wray L, June CH, Maude SL, Frey NV, Grupp SA. CD22-targeted chimeric antigen receptor-modified T cells for children and adults with relapse of B-cell acute lymphoblastic leukemia after CD19-directed immunotherapy. J Immunother Cancer. 2025 Apr 17;13(4):e011549. doi: 10.1136/jitc-2025-011549. PMID 40246579
- [Derived] Singh N, Frey NV, Engels B, Barrett DM, Shestova O, Ravikumar P, Cummins KD, Lee YG, Pajarillo R, Chun I, Shyu A, Highfill SL, Price A, Zhao L, Peng L, Granda B, Ramones M, Lu XM, Christian DA, Perazzelli J, Lacey SF, Roy NH, Burkhardt JK, Colomb F, Damra M, Abdel-Mohsen M, Liu T, Liu D, Standley DM, Young RM, Brogdon JL, Grupp SA, June CH, Maude SL, Gill S, Ruella M. Antigen-independent activation enhances the efficacy of 4-1BB-costimulated CD22 CAR T cells. Nat Med. 2021 May;27(5):842-850. doi: 10.1038/s41591-021-01326-5. Epub 2021 Apr 22. PMID 33888899